CLINICAL TRIAL: NCT06164834
Title: A Randomized, Open-label, Three-period, Multiple Dosing Crossover Clinical Trial to Evaluate the Influence of Tegoprazan on the Pharmacodynamics of Clopidogrel in Healthy Subjects
Brief Title: Effect of Tegoprazan on Pharmacodynamics of Clopidogrel in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_123
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel; tegoprazan; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clopidogrel 75 mg (Active Comparator): Oral administration of clopidogrel 75 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75 mg
- Clopidogrel 75 mg + Tegoprazan 25 mg (Experimental): Oral administration of clopidogrel 75 mg tablet and tegoprazan 25 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75 mg; Drug: Tegoprazan 25 mg
- Clopidogrel 75 mg + Esomeprazole 20 mg (Experimental): Oral administration of clopidogrel 75 mg tablet and esomeprazole 20 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75 mg; Drug: Esomeprazole 20mg

INTERVENTIONS:
Drug: Clopidogrel 75 mg — Clopidogrel 75 mg tablet
  Other Names: Plavix
Drug: Tegoprazan 25 mg — Tegoprazan 25 mg tablet
  Other Names: K-CAB
  Arms: Clopidogrel 75 mg + Tegoprazan 25 mg
Drug: Esomeprazole 20mg — Esomeprazole 20 mg tablet
  Other Names: Nexium
  Arms: Clopidogrel 75 mg + Esomeprazole 20 mg

SUMMARY:
This study aims to evaluate the effects of tegoprazan or esomeprazole administered in combination with clopidogrel on the pharmacodynamics/Pharmacokinetics of clopidogrel in healthy adults

DETAILED DESCRIPTION:
Evaluation Criteria:

* Primary outcome Pharmacodynamic assessments using P2Y12 assay
* Secondary outcome Pharmacokinetics assessments on Cmax,ss, Cmin,ss, Cavg,ss, AUCτ,ss, Tmax,ss, t1/2,ss, CLss/F, Vd,ss/F, and PTF of clopidogrel
* Safety assessments with adverse event monitoring including subjective/ objective symptoms, physical examination, vital signs, electrocardiogram, and laboratory test

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 years and ≤ 50 years on the date of the written informed consent
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2 at the time of screening
* Is given a detailed explanation and fully understood the study, then voluntarily decided to participate and provided written informed consent before any screening procedure
* Negative for serum Helicobacter pylori antibodies
* Judged by the investigator to be eligible for this study based on physical examination, laboratory test, inquiry, etc.

Exclusion Criteria:

* Presence or history of clinically significant liver, kidney, nervous system, respiratory system, endocrine system, blood and tumor, cardiovascular system, urinary system or psychiatric disease
* Presence or history of gastrointestinal disorder (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux disease, Crohn's disease, etc.) that may influence the safety and pharmacodynamic assessments of the investigational product and history of gastrointestinal surgery (except simple appendectomy and hernia surgery), hemostatic disorder or hemorrhage-related disease
* Hypersensitivity to drugs including the ingredients of the investigational product and other drugs (aspirin, antibiotics, etc.) or history of clinically significant hypersensitivity
* Positive result in serology tests (Hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test)
* Blood total bilirubin, AST (GOT), and ALT (GPT) > 1.5 x upper limit of normal range at the screening test
* Platelet, PT and aPTT levels outside the upper/lower limit of normal range by 10% at the screening test
* Systolic blood pressure is < 90 mmHg or > 139 mmHg, diastolic blood pressure < 50 mmHg or > 89 mmHg, or pulse rate is < 45 beats/minute or > 100 beats/minute when vital signs are measured in sitting position after resting for at least 3 minutes at the screening test
* Showing the following findings on ECG at the screening test: QTc > 450 msec, PR interval > 210 msec, QRS interval > 120 msec, Other clinically significant findings
* P2Y12 Reaction Unit (PRU) outside the upper/lower limit of normal range by 10% as a result of P2Y12 assay at the screening test
* History of drug abuse or positive urine screening for drug abuse
* Considered ineligible to participate in the study by the investigator based on laboratory test results or other reasons

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-05 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in P2Y12 Reaction Unit (PRU) from baseline | Pre-dose(0h) on days 1, 3, 5, 7 and 8 in each period
  Pharmacodynamic blood sampling to measure PRU using VerifyNow® system

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hwan Lee, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea